CLINICAL TRIAL: NCT01167088
Title: A Double-blind Randomised Placebo-controlled Multicentre Study of 40mg MitoQ and Placebo for the Treatment of Participants With Raised Liver Enzymes Due to Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: A Study to Compare MitoQ and Placebo to Treat Non-alcoholic Fatty Liver Disease (NAFLD)
Acronym: MARVEL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated due to poor participant recruitment
Sponsor: Antipodean Pharmaceuticals, Inc. (Industry)
Responsible Party: Dr Ken Taylor, CEO, Antipodean Pharmaceuticals Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTQ-LD-001; 2010-021368-13 (EudraCT Number)
Record Dates: First submitted 2010-07-19; First posted 2010-07-22 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Double-blind; Placebo-controlled; Non-alcoholic fatty liver disease; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mitoquinone mesylate tablets (MitoQ) (Experimental)
  Interventions: Drug: Mitoquinone mesylate
- Matching placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mitoquinone mesylate — 2 tablets to be taken daily upon wakening, with a glass of water and at least one hour before food.
  Arms: Mitoquinone mesylate tablets (MitoQ)
Drug: Placebo — Placebo
  Arms: Matching placebo tablet

SUMMARY:
The purpose of this study is to investigate whether a new medicine, called mitoquinone, will reduce raised liver enzymes due to NAFLD and to see if it is safe.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. NAFLD as determined by raised ALT (> 1.5 x ULN corresponding to >29U/L for females and >45U/L for males] in the screening period and on at least two other occasions in the previous 6 months) and ultrasound evidence of steatosis (in the previous 12 months).
3. Be aged between 18 - 70 years on the day of consent
4. Expect to not require or make any changes in all their current concomitant medications (prescribed and over-the-counter) for the duration of their participation in the study
5. Female patients with reproductive potential must have a negative serum pregnancy test within 14 days prior to start of trial and must agree to use a medically acceptable method of contraception throughout the treatment period and for 1 month after discontinuation of treatment. Acceptable methods of contraception include IUD, oral contraceptive, subdermal implant and double barrier (condom with a contraceptive sponge or contraceptive pessary)

Exclusion Criteria:

1. Alcohol consumption > 14 units/week for females and 21 units/week for males
2. Hepatocellular carcinoma (HCC) or suspicion of HCC
3. Presence of human immunodeficiency virus (HIV), Hepatitis B (HBV) or Hepatitis C (HCV)
4. Renal impairment (creatinine > 1.5 x ULN) or hepatorenal syndrome
5. Chronic pancreatitis
6. Hospitalization for liver disease within 60 days of the baseline visit
7. Previously diagnosed diabetes / treatment with insulin sensitizing agents
8. Severe or morbid obesity (BMI>40kg/m2)
9. ALT or AST > 10 times ULN
10. Liver transplant recipients
11. Corticosteroids in the past 30 days
12. Any participant who has received any investigational drug or device within 30 days of dosing, or who is scheduled to receive another investigational drug or device during the course of this trial
13. A history of a malignancy other than treated basal cell or squamous cell carcinoma of the skin; those with a history of malignancy that has been treated with no recurrence within the last 2 years are not excluded
14. Females who are pregnant or breastfeeding
15. Use of Coenzyme Q10, either prescribed or purchased over-the-counter, are prohibited during the study, except for doses of up to 25mg/day which have been stable for 30 days prior to baseline. Higher doses require a 7 day washout prior to baseline.
16. Use of Vitamin E, either prescribed or purchased over-the-counter, are prohibited during the study, except for doses of up to 200IU/day which have been stable for 30 days prior to baseline. Higher doses require a 90 day washout prior to baseline.
17. Any changes to prescription medication in the 30 days prior to baseline
18. A history of a hypersensitivity reaction to any components of the study drug or structurally similar compounds including Coenzyme Q10 and idebenone
19. Unable to swallow tablets whole
20. Patients with histological or clinical evidence of established cirrhosis
21. Suffering from any other disease or condition which, in the opinion of the investigator, means that it would not be in the patient's best interest to participate in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Percentage change in ALT (relative to baseline) at the end of the treatment period (Day 90) for MitoQ compared with placebo. | Baseline and 3 months

SECONDARY OUTCOMES:
Absolute change in ALT level (relative to baseline) at end of treatment period for MitoQ compared with placebo | Baseline and 3 months
The percentage of participants whose ALT levels are in the normal range at the end of the treatment period. | 3 months
The difference in the percentage and absolute rates of change in ALT levels between MitoQ and placebo. | Baseline to 3 months
The percentage and absolute change in AST at the end of the treatment period (relative to baseline) for MitoQ compared with placebo. | Baseline and 3 months
The change in HOMA-IR at the end of the treatment period (relative to baseline) for MitoQ compared with placebo. | Baseline and 3 months
The change in HbA1c at the end of the treatment period (relative to baseline) for MitoQ compared with placebo. | Baseline and 3 months
The percentage and absolute change in GGT and alkaline phosphatase at the end of the treatment period (relative to baseline) for MitoQ compared with placebo. | Baseline and 3 months
Areas under the ALT, AST, GGT and alkaline phosphatase curves from baseline to the end of the treatment period. | Baseline to 3 months
The change in markers of liver inflammation (leptin and adiponectin) at the end of the treatment period (relative to baseline) for MitoQ compared with placebo. | Baseline and 3 months
The change in biomarkers of mitochondrial function and oxidative damage (isoprostanes) at the end of the treatment period (relative to baseline) for MitoQ compared with placebo. | Baseline and 3 months
The change in blood pressure at the end of the treatment period (relative to baseline) for MitoQ compared with placebo. | Baseline and 3 months
The change in blood lipid profile at the end of the treatment period (relative to baseline) for MitoQ compared with placebo. | Baseline and 3 months
Incidence of adverse events | Baseline to Follow-up (total 4 months)
Clinically relevant deterioration in laboratory variables | Baseline to Follow-up (total 4 months)
Clinically relevant deterioration in vital signs | Baseline to Follow-up (total 4 months)
Clinically relevant deterioration in ECG parameters | Baseline to Follow-up (total 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Day, MD, PhD, Principal Investigator — Newcastle University Medical School, UK
Locations (1):
- Freeman Hospital, Newcastle upon Tyne, United Kingdom